CLINICAL TRIAL: NCT04009421
Title: Covariates of Coronary Artery Plaque Burden and Composition by CT Coronary Angiography in Women and Men With Stable Angina and Non-obstructive Coronary Artery Disease - Analysis From the NORIC Registry
Brief Title: Coronary Artery Plaque Burden in Stable Angina and Non-obstructive Coronary Artery Disease
Status: Active, not recruiting | Type: Observational
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Mai Tone Lønnebakken, Professor, University of Bergen
Other Study IDs: 1573
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease; Plaque, Atherosclerotic
Keywords: coronary artery disease; plaque burden; prognosis
MeSH Terms: conditions — Coronary Artery Disease; Plaque, Atherosclerotic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High and low coronary artery plaque burden: Patients with high plaque burden defined as plaque in >=4 segments of the coronary tree and low plaque burden as plaque in <4 segments of the coronary tree assessed by postprocessing of CT coronary angiography images and cardiovascular events and mortality.
  Interventions: Diagnostic Test: Coronary artery plaque assessment by CT coronary angiography QAngio CT RE

INTERVENTIONS:
Diagnostic Test: Coronary artery plaque assessment by CT coronary angiography QAngio CT RE — Assessment of segmental plaque volume and composition

SUMMARY:
Non-obstructive coronary artery disease (CAD), particularly common in women, has been associated with impaired quality of life and risk of recurrent hospitalizations. Several studies have also demonstrated increased risk of incident acute coronary events and mortality.

The main objective of the project is to assess the association between coronary artery plaque features by coronary CT angiography and long term prognosis in a large unselected population undergoing CT coronary angiography due to stable angina and suspected myocardial ischemia from the Norwegian Registry for Invasive Cardiology (NORIC) diagnosed with non-obstructive CAD by coronary CT angiography.

DETAILED DESCRIPTION:
Patients with stable angina and non-obstructive coronary artery disease by CT coronary angiography will be selected from the Norwegian Registry of Invasive Cardiology (NORIC). This is a national quality control registry run and controlled by the Norwegian Institute of Public Health (www.fhi.no). All CT coronary angiograms will be reanalyzed using advanced post-processing analysis software to assess coronary artery plaque burden, distribution and composition. Through linking with the Norwegian Cardiovascular Disease Registry and the Cause of Death Registry (www.fhi.no) we will be able to assess the association between long-term prognosis (5 years) and coronary artery plaque features.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina
* Non-obstructive coronary artery disease by CT coronary angiography defined as <50% stenosis (lumen diameter reduction)

Exclusion Criteria:

* Obstructive coronary artery disease
* Unstable angina
* Previous myocardial infarction, heart surgery or percutaneous coronary interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from the NORIC registry undergoing CT coronary angiography due to chest pain and suspected myocardial ischemia and diagnosed with non-obstructive coronary artery disease between 2013-2017.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular mortality and nonfatal acute myocardial infarction | 5 years
  Composite of deaths caused by cardiovascular disease and nonfatal acute myocardial infarction

SECONDARY OUTCOMES:
All-cause mortality, hospitalization due to cardiovascular disease and revascularization procedures | 5 years
  All-cause mortality, hospitalization due to cardiovascular disease and revascularization procedures

CONTACTS AND LOCATIONS:
Overall Officials: Mai Tone Lønnebakken, MD phd, Principal Investigator — University of Bergen
Locations (1):
- Department of Clinical Science, University of Bergen, Bergen, Norway

REFERENCES:
- [Derived] Hondros CAB, Hanseth S, Solvik M, Pedersen EKR, Khan I, Hovland S, Larsen TH, Lonnebakken MT. Age-stratified differences in coronary artery plaque phenotypes in women and men with non-obstructive coronary artery disease. Open Heart. 2025 Jul 11;12(2):e003371. doi: 10.1136/openhrt-2025-003371. PMID 40645670
- [Derived] Khan I, Hondros CAB, Hanseth S, Pedersen ER, Hovland S, Larsen TH, Lonnebakken MT. Epicardial adipose tissue volume, compositional plaque progression, and vulnerability in nonobstructive coronary artery disease. Coron Artery Dis. 2025 Nov 1;36(7):580-586. doi: 10.1097/MCA.0000000000001539. Epub 2025 Jun 17. PMID 40521640
- [Derived] Hondros CAB, Khan I, Solvik M, Hanseth S, Pedersen EKR, Hovland S, Larsen TH, Lonnebakken MT. Compositional plaque progression in women and men with non-obstructive coronary artery disease. Int J Cardiol Heart Vasc. 2024 Feb 7;51:101352. doi: 10.1016/j.ijcha.2024.101352. eCollection 2024 Apr. PMID 38356931
- [Derived] Berge CA, Eskerud I, Almeland EB, Larsen TH, Pedersen ER, Rotevatn S, Lonnebakken MT. Relationship between hypertension and non-obstructive coronary artery disease in chronic coronary syndrome (the NORIC registry). PLoS One. 2022 Jan 21;17(1):e0262290. doi: 10.1371/journal.pone.0262290. eCollection 2022. PMID 35061769